CLINICAL TRIAL: NCT04045535
Title: Effectiveness of a Physical Activity Intervention in the Quality of Life of Pre-frail Older Adults Aged 65 Years or Over With Chronic Pain. Randomized Controlled, Multicenter and Pragmatic Trial in Primary Care.
Brief Title: Effectiveness of a Physical Activity Intervention for Pre-frail Older Adults With Chronic Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gerencia de Atención Primaria, Madrid (Other Government)
Responsible Party: Principal Investigator, Pedro Otones Reyes, Principal Investigator. Cinical nurse, Gerencia de Atención Primaria, Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT180719
Record Dates: First submitted 2019-07-30; First posted 2019-08-05 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Frailty; Chronic Pain; Old Age; Debility
Keywords: Primary Health Care; Nursing Intervention; Physical Activity
MeSH Terms: conditions — Frailty; Chronic Pain; Motor Activity

STUDY DESIGN:
Masking Description: Intervention can't be masked. Statistician conducting the analysis will not know to which study arm a given patient has been assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention with nurse and patients
  Interventions: Other: Physical Activity Program; Other: Usual care
- Usual care (Active Comparator): Usual clinical care based on current clinical practice guidelines.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Physical Activity Program — Usual Care and a nurse-led physical activity program once a week for 8 weeks. Each session last for 60 minutes, 15 for warming-up and 45 for different exercises.
  Arms: Intervention group
Other: Usual care — Usual clinical care based on current clinical practice guidelines.

SUMMARY:
The purpose of this investigation is to evaluate the effectiveness of a multicomponent structured physical exercise program for adults aged 65 years or more, classified as pre-frail and with chronic pain to improve the Perceived Health Related Quality of Life, compared with usual care.

DETAILED DESCRIPTION:
Design: Randomized controlled, pragmatic clinical trial with two groups and 3 months follow-up.

Unit of randomization: Patient. Unit of analysis: Patient. Setting: A Primary Health Care Center in the Spanish Autonomous Community of Madrid.

Population: Pre-frail patients aged 65 years or more with chronic pain. Intervention: Multicomponent structured physical exercise program. Control group: Usual care. Variables: Perceived Health Related Quality of Life (EuroQol 5D-5L), Pain Intensity (Visual Analogue Scale), Frailty (SHARE-Frailty Index), Physical Performance (Short Physical Performance Battery, SPPB), Depression (Yesavage).

Analysis: Mean change differences after 3 months in EQ5D dimensions between groups with CI 95%. Mean differences or proportion differences will be calculated according to variable characteristics between groups with appropriate statistical test.

ELIGIBILITY:
Inclusion Criteria:

* Clinical record of Chronic Pain by International Classification of Primary Care (ICPC) Code A01.
* Being classified as pre-frail by SHARE-FI questionnaire.
* Informed consent

Exclusion Criteria:

* Housebound patients
* Institutionalized patients
* Not living in the area of the investigation
* Dependence for bADL
* Not being fluent in Spanish
* Severe mental illness or cognitive disorder

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-07-02 (Actual)

PRIMARY OUTCOMES:
Perceived Health Related Quality of Life | Change from baseline at 2 and 5 months
  Quality of life assessed by EuroQol 5 Dimen (EQ5D-5L) Scale. It consist on a Quality Index (Range 0-1) calculated from scores of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) with value for Spain set and a Visual Analog Scale (Range 0: Worst possible health-100: Best possible health).

SECONDARY OUTCOMES:
Pain Intensity | Change from baseline at 2 and 5 months
  Pain Intensity was assessed by McGill Pain Questionnaire's Visual Analog Scale (VAS). It consists on a 100mm horizontal line in which patient points the intensity of his pain. It is measured from left to right. Left side of the line (0 millimeters, mm) means "no pain" and it is the minimum score and right side of the line (100mm) means "pain as worst as you can imagine" and it is maximum score. Lower punctuation meana better outcomes.
Frailty Status | Change from baseline at 2 and 5 months
  Frailty Status assessed by SHARE-FI (Survey of Health, Ageing and Retirement Frailty Index). It consists on summarizing the response to 5 criteria (exhaustion, weight loss, weakness, slowness and low active) in a discreet factor (DFS). Scores are different for men and women.
  Women: If predicted DFS < 0.31, NON-FRAIL; If predicted DFS < 2.13, PRE-FRAIL; If predicted DFS < 6, FRAIL Men: If predicted DFS < 1.21, NON-FRAIL; If predicted DFS < 3.00, PRE-FRAIL; If predicted DFS < 7, FRAIL
Physical Performance | Change from baseline at 2 and 5 months
  Assessed by Short Physical Performance Battery (SPPB). It evaluates balance, walk speed and sitting and standing in a chair. Each Item is scored 0-4 points. Yielding a total between 0 (worst physical performance ) and 12 (best physical performance).
Falls | At 2 months and at 5 months
  Number of falls during the follow-up process
Depression | Change from baseline at 2 and 5 months
  Assessed by ultra-short Yesavage Scale (Geriatric Depression Scale, GDS-5). It consist on 5 questions of the GDS-15 questionnaire (Range:0-5. Cutpoint for depression: 2).
Basic Activities of Daily Living (bADL) | Change from baseline at 2 and 5 months
  Assessed by Barthel Scale. It assesses the help needed with ten variables: feeding, bathing, grooming, dressing, urinary incontinence, faecal incontinence, toilet use, transfers bed to chair, mobility and climbing stairs. (Range: 0: Full Dependence - 100: Independence for bADL).
Number of meetings attended | At 2 months
  Number of meetings attended by the participants from intervention group.
Satisfaction with the intervention | At 2 months
  Assessed with Client Satisfaction Questionnaire (CSQ-8). It consist on 8 questions (four ranged 4: most satisfaction-1: least satisfaction and four ranged 1: most satisfaction -4 least satisfaction)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Otones Reyes, RN, PhDc, Principal Investigator — Gerencia de Atención Primaria, Madrid; Eva García Perea, RN, PhD, Study Director — Universidad Autonoma de Madrid; Azucena Pedraz Marcos, RN, PhD, Study Director — Universidad Autonoma de Madrid
Locations (1):
- Gerencia de Atención Primaria, Madrid, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Otones P, Garcia E, Sanz T, Pedraz A. A physical activity program versus usual care in the management of quality of life for pre-frail older adults with chronic pain: randomized controlled trial. BMC Geriatr. 2020 Oct 8;20(1):396. doi: 10.1186/s12877-020-01805-3. PMID 33032532